CLINICAL TRIAL: NCT01989858
Title: ITACA-S2(Intergroup Trial in Adjuvant Chemotherapy for Adenocarcinoma of the Stomach:Comparison of the Efficacy of a Peri-operative Versus a Post-operative Chemotherapy Treatment in Patients With Operable Gastric Cancer and Assessment of the Benefit of a Post-operative Chemo-radiotherapy.
Brief Title: ITACA-S2 (Intergroup Trial in Adjuvant Chemotherapy for Adenocarcinoma of the Stomach)
Acronym: ITACA-S2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of clinical cases
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021052-25
Record Dates: First submitted 2011-06-16; First posted 2013-11-21 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2010-07

CONDITIONS: Gastric Adenocarcinoma
Keywords: localized gastric adenocarcinoma, operable considered.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- peri-operative CHT (Arm A) (Experimental): In peri-operative CHT arm CHT will be administered within 1 week (+3 days) after randomization, surgery will be performed after re-staging and 3+1 weeks after completion of the third cycle of CHT (approximately 13+1 weeks after randomization). Then CHT will be re-administered 5+1 weeks after surgery.
  Interventions: Other: peri-operative cht
- post-operative CHT (Arm B) (Active Comparator): In post-operative CHT arm, surgery will take place 3+1 weeks after randomization and CHT will be administered 5+1 weeks after surgery (approximately 8+1 weeks after randomization).
  Interventions: Other: post-operative CHT
- peri-operative CHT + post-operative CHT-RTX (Arm C) (Experimental): CHT 1 week (+3 days) after randomization surgery after re-staging and 3+1 weeks after completion of the third cycle of CHT CHT 5+1 weeks after surgery.
  Interventions: Other: peri-operative cht + post-operative cht-rtx
- post-operative CHT + post-operative CHT-RTX (Arm D) (Active Comparator): surgery will take place 3+1 weeks after randomization and CHT will be administered 5+1 weeks after surgery (approximately 8+1 weeks after randomization).
  Interventions: Other: post-operative cht + post-operative cht-rtx

INTERVENTIONS:
Other: peri-operative cht — CHT treatment have to be chosen between the following associations:
  Chemotherapy regimen containing epirubicin, cisplatin and capecitabine (EOX) E: epirubicin 50 mg/m² intravenous (iv) bolus, day 1 every 3 weeks O: oxaliplatin 130 mg/m² iv infusion, day 1 in 2-3 hours every 3 weeks X: capecitabine 625 mg/m² bis in die (bid), day 1 per os (po) continuously
  or
  Chemotherapy regimen containing epirubicin, cisplatin and 5-fluorouracil (ECF) E: epirubicin 50 mg/m² iv bolus, day 1 every 3 weeks C: cisplatin 60 mg/m² iv with standard hydration day 1 every 3 weeks F: 5FU 200 mg/m² daily by continuous infusion via central line.
  Arms: peri-operative CHT (Arm A)
Other: post-operative CHT — CHT treatment have to be chosen between the following associations:
  EOX E: epirubicin 50 mg/m² intravenous (iv) bolus, day 1 every 3 weeks O: oxaliplatin 130 mg/m² iv infusion, day 1 in 2-3 hours every 3 weeks X: capecitabine 625 mg/m² bis in die (bid), day 1 per os (po) continuously
  or ECF E: epirubicin 50 mg/m² iv bolus, day 1 every 3 weeks C: cisplatin 60 mg/m² iv with standard hydration day 1 every 3 weeks F: 5fluorouracil (5FU) 200 mg/m² daily by continuous infusion via central line.
  Arms: post-operative CHT (Arm B)
Other: peri-operative cht + post-operative cht-rtx — CHT treatment have to be chosen between the following associations:
  * EOX E: epirubicin 50 mg/m² intravenous (iv) bolus, day 1 every 3 weeks O: oxaliplatin 130 mg/m² iv infusion, day 1 in 2-3 hours every 3 weeks X: capecitabine 625 mg/m² bis in die (bid), day 1 per os (po) continuously or
  * ECF E: epirubicin 50 mg/m² iv bolus, day 1 every 3 weeks C: cisplatin 60 mg/m² iv with standard hydration day 1 every 3 weeks F: 5FU 200 mg/m² daily by continuous infusion via central line.
  The prescribed RTX dose to clinical target volume should be 45 gray (Gy) delivered in daily fraction of 1.8 Gy, five times per week for six weeks. RTX will be administered concurrently with CHT. The choice of the associated CHT should be between the following schedules:
  * 5FU 225 mg/m² given as a continuous iv infusion or
  * capecitabine 825 mg/m² bid given as a continuous oral administration during the entire course of RTX.
  Arms: peri-operative CHT + post-operative CHT-RTX (Arm C)
Other: post-operative cht + post-operative cht-rtx — CHT treatment have to be chosen between the following associations:
  * EOX E: epirubicin 50 mg/m² intravenous (iv) bolus, day 1 every 3 weeks O: oxaliplatin 130 mg/m² iv infusion, day 1 in 2-3 hours every 3 weeks X: capecitabine 625 mg/m² bis in die (bid), day 1 per os (po) continuously or
  * ECF E: epirubicin 50 mg/m² iv bolus, day 1 every 3 weeks C: cisplatin 60 mg/m² iv with standard hydration day 1 every 3 weeks F: 5FU 200 mg/m² daily by continuous infusion via central line.
  The prescribed RTX dose to clinical target volume should be 45 gray (Gy) delivered in daily fraction of 1.8 Gy, five times per week for six weeks. RTX will be administered concurrently with CHT. The choice of the associated CHT should be between the following schedules:
  * 5FU 225 mg/m² given as a continuous iv infusion or
  * capecitabine 825 mg/m² bid given as a continuous oral administration during the entire course of RTX.
  Arms: post-operative CHT + post-operative CHT-RTX (Arm D)

SUMMARY:
The study addresses two primary questions, according to its factorial design:

* to compare the efficacy in terms of overall survival (OS) of a peri-operative vs. a post-operative chemotherapy (CHT) treatment, irrespectively of the presence of a post-surgical chemo-radiotherapy (CHT-RTX) (Timing Study);
* to compare the efficacy in terms of relapse free survival (l-RFS) of a post-surgical CHT-RTX treatment vs. no other treatment, irrespectively of the timing of CHT (RTX Study).

The study has a 2x2 factorial design, thus consisting of two independent, following specific eligibility criteria and with different randomization scheme studies, the Timing Study and the RTX Study.

Both studies are Italian, multicentre, open-label, randomized, superiority, phase III trials conducted in patients with histologically confirmed, localized gastric adenocarcinoma, which is considered operable.

In the Timing Study patients fulfilling the eligibility criteria will be randomized with a 1:1 ratio to receive:

* peri-operative CHT (Arm A) or
* post-operative CHT (Arm B) Once randomized in the Timing Study, patients may also be randomized in the RTX

Study to receive in addition to CHT a post-operative CHT-RTX treatment or no other treatment. This is possible since the randomization will be done in two steps: the first for the Timing Study for all the participating centres (peri-operative CHT vs. post-operative CHT) and the second one for the RTX Study, only for those centres with the radiotherapist willing and able to participate (post- surgical CHT-RTX vs. no other treatment). Thus the following four arms will be generated:

* peri-operative CHT (Arm A)
* post-operative CHT (Arm B)
* peri-operative CHT + post-operative CHT-RTX (Arm C)
* post-operative CHT + post-operative CHT-RTX (Arm D) The study will be conducted in more than one hundred experimental centres. Follow-up F(-up) procedures and timing of the visits will be consistent with current clinical practice.

Based on case-mix of sample 1000-1180 patients are needed in the Timing study and 420-520 in the RTX study.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* Eastern Cooperative Oncology Group - Performance Status (ECOG-PS) 0-1
* T3 or T4 carcinoma without lymphnode involvement (N0) and any T-stage with (N+) lymphnode involvement
* no distant metastases (M0)
* fitness to receive CHT and CHT-RTX
* no peripheral neuropathy greater than grade 1
* absence of peritoneal carcinomatosis
* written informed consents (one for each trial) given before the randomization, according to International Conference on Harmonisation/Good Clinical Practice (ICH/GCP)

Exclusion Criteria:

* adenocarcinoma of the gastro-esophageal junction
* previous CHT or RTX
* abnormal haematological, hepatic or renal functions, assessed within 7 days prior to randomization
* lymphnode metastases (biopsy proof, if possible) outside the loco-regional field, such as supraclavicular, mediastinal or para-aortic nodes
* positive peritoneal cytology
* clinical significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤ 6 months), myocardial infarction (≤ 6 months), instable angina, New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication
* history or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or patients at high risk from treatment complications
* pregnancy or breast feeding. Women of childbearing potential and their parents must be willing to practice acceptable methods of birth control to prevent pregnancy
* presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and f-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS)- Timing Study | 5 years
  OS, defined for each patient as the time from the date of randomization to the date of death from any cause. Patients not reported as having died at the end of the study will be censored at the date they were last known to be alive.

SECONDARY OUTCOMES:
Dose-intensity | up to 8 weeks
  * Dose-intensity, that is the dose of effective drug administrated per unit time (mg/m2/week or Gy/week)
  * Dose and/or time modifications
  * Premature withdrawals
Maximum toxicity grade | up to 8 weeks
  * Maximum toxicity grade experienced by each patient for each toxicity
  * Patients experiencing grade 3-4 toxicity for each toxicity
  * Type,frequency and nature of serious adverse events (SAEs)
  * Patients with at least a SAE
  * Patients with at least a serious adverse drug reaction (SADR)
Disease Free Survival (DFS) - Timing Study | 3 years
  DFS, defined for each patient as the time from the date of randomization to the date of local or regional relapse, distant metastasis, second primary malignancy or death from any cause, whichever comes first. Patients not recurred, progressed or died while on study or lost to f-up will be censored at their last disease assessment date.
Relapse Free Survival (l-RFS)- RTX Study | 3 years
  1-RFS, defined for each patient as the time from the date of randomization to the date of first local recurrence or death from any cause, whichever comes first.
  Description: 1-RFS, defined for each patient as the time from the date of randomization to the date of first local recurrence or death from any cause, whichever comes first. Patients not locally recurred or died while on study or lost to f-up will be censored at their last disease assessment date

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Di Costanzo, MD, Principal Investigator — Azienda Ospedaliero- Universitaria Careggi - Firenze U.O. Medica
Locations (32):
- Italy (32):
  - Ospedali Riuniti di Bergamo, Bergamo, BG
  - A. O. Ospedale Treviglio-Caravaggio, Treviglio, BG
  - A.O. Sant'Orsola Malpighi, Bologna, BO
  - Policlinico Sant'Orsola Malpighi, Bologna, BO
  - A.O. Santa Croce e Carle, Cuneo, CN
  - Azienda Ospedaliero-Universitaria "Policlinico-Vittorio Emanuele", Catania, CT
  - Policlinico Universitario Mater Domini, Catanzaro, CZ
  - Azienda Ospedaliero- Universitaria Careggi - Firenze, Florence, FI
  - A.O. Ospedale San Gerardo, Monza, MB
  - Azienda Ospedaliera di Desio e Vimercate, Vimercate, MB
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Milan, MI
  - Istituto Nazionale per la Cura e lo Studio dei Tumori, Milan, MI
  - Istituto Oncologico Europeo, Milan, MI
  - Azienda Ospedaliera "San Paolo", Milan, MI
  - Istituto Clinico Humanitas, Rozzano, MI
  - Casa di Cura MultiMedica, Sesto San Giovanni, MI
  - A. O. "Carlo Poma", Mantova, MN
  - Ospedale "Ramazzini " di Carpi, Carpi, MO
  - Ospedale "Guglielmo da Saliceto", Piacenza, PC
  - IRCCS Istituto Oncologico Veneto, Padua, PD
  - Ospedale Misericordia e Dolce - USL 4, Prato, PO
  - Ospedale Santa Croce Fano, Fano, PU
  - Azienda Ospedaliera 'San Carlo', Potenza, PZ
  - Arcispedale S. Maria Nuova Azienda Ospedaliera, Reggio Emilia, RE
  - Università "Campus Bio-Medico", Roma, RM
  - Policlinico Universitario A. Gemelli, Roma, RM
  - A.O. della Valtellina e della Valchiavenna - "Ospedale E. Morelli", Sondalo, SO
  - IRCC/FPO -Istituto per la Ricerca e la Cura del Cancro di Candiolo, Candiolo, TO
  - A. O. "Ospedale di Circolo di Busto Arsizio" - Busto Arsizio (VA), Busto Arsizio, VA
  - A. O. Busto Arsizio - P.O. Saronno, Saronno, VA
  - A.O. Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Fondazione "G. Pascale" Istituto Tumori di Napoli, Napoli